CLINICAL TRIAL: NCT02217046
Title: Phase 1 Study of Prevention of Cardiac Device Replacement Site Infection
Brief Title: Decrease Implantation Site INFECTION : a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, Ph.D, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DISINFECTION II
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Infection
Keywords: Infection; prevention; cardiac devices
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- device replacement (Experimental): remove previously inserted cardiac device and posterior pocket capsule. the pocket that will receive the heart mechanism is sterilized with a hydroperoxide soaked gauze
  Interventions: Procedure: device replacement(pocket capsule removal)
- control group (No Intervention): remove previously inserted cardiac device and the pocket that will receive the heart mechanism is sterilized with a hydroperoxide soaked gauze

INTERVENTIONS:
Procedure: device replacement(pocket capsule removal) — remove previously inserted cardiac device and posterior pocket capsule. the pocket that will receive the heart mechanism is sterilized with a hydroperoxide soaked gauze
  Arms: device replacement

SUMMARY:
Cardiovascular implantable electronic device (CIED) infections have been increasing out of proportion to the number of devices implanted the investigators investigated recent trends and possible causes of the increasing numbers of Cardiovascular implantable electronic device infections.

DETAILED DESCRIPTION:
There are many studies on the preventive use of Antibiotics or povidone iodine to Cardiovascular implantable electronic device (CIED) infections.

But, studies of posterior pocket capsule removal is still limited.

The investigators had planned research on effects of posterior pocket capsule removal before cardiac devices replacement.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cardiac devices replacement

Exclusion Criteria:

* under the age of 18
* take an antibiotic
* history of infection within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2013-12; Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
freedom of cardiac device-related infection | 1 year after precedure
  check the symptoms of infection. If have symptoms of infection : check the fever, heart rate, respiration rate, blood test, EKG

SECONDARY OUTCOMES:
freedom of endocarditis | 1 year after precedure
  check the symptoms of infection. If have symptoms of infection : check the fever, heart rate, respiration rate, blood test, EKG

OTHER OUTCOMES:
freedom of general infection | 1 year after procedure
  check the symptoms of infection. If have symptoms of infection : check the fever, heart rate, respiration rate, blood test, EKG

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seog Oh, Ph.D, Study Chair — Seoul St. Mary's Hospital
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Ch-gu, South Korea